CLINICAL TRIAL: NCT02911038
Title: Stereolithographic Technique for Complete Denture Fabrication
Brief Title: Stereolithographic Technique for Dentures
Acronym: PRIDENTPRO
Status: Completed | Type: Observational
Sponsor: Corina Marilena Cristache (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); Romanian National Authority for Scientific Research and Innovation (UEFISCIDI) (Unknown); University Politechnica of Bucharest (Unknown); TURKEY MEDISEN Ltd (Unknown); DDX Europa SRL, Bucharest, Romania (Unknown)
Responsible Party: Sponsor-Investigator, Corina Marilena Cristache, Senior Lecturer, PhD, Dr, Concordia Dent Srl
Organization: Concordia Dent Srl (Other)
Other Study IDs: CCDI-UEFISCDI 30/2016
Record Dates: First submitted 2016-09-18; First posted 2016-09-22 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Mouth Edentulous; Jaw Edentulous
Keywords: Complete denture; PMMA; Stereolithography
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this observational study is: producing complete dental prosthesis with the aid of CAD-CAM (Computer aided design & manufacturing) - 3D printing (Stereolithography) technology - using as printable material Poli(methylmetacrylate) - PMMA - with Nano TiO2 nanoparticles composite completely characterized.

DETAILED DESCRIPTION:
In order to improve complete dentures fabrications an experimental model for optimizing the composite material and the execution technique for the 3D printed dental prosthesis was developed.

* A new polymer - nano-TiO2 composite system for dentures printing was obtained by adding 0,4-1%TiO2 nanoparticle in the commercially available E-Dent 100 (EnvisionTEC, Germany).
* The new polymer was completely characterized and biocompatibility tests were perform.
* A stereolithography technique was set-up for CAD-CAM complete dentures manufacturing.
* 3D printed dental prosthesis will be inserted to a number of 35 complete edentulous patients from a target group;
* Clinical follow-up at 6, 12 and 18 months and quality assessment of the dentures will be recorded in a specific chart.
* A statistical evaluation of data recorded during the entire follow-up period will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mobile or removable dentures after establishing diagnosis and treatment plan, following initial clinical and laboratory examinations,
* Persons having mental competence, decision-making capacity, legal competence.
* Patients willing to accept complete denture treatment.
* Patients with good systemic health, able to attend all the follow-up sessions.
* Patients accepting the participation in the study, including the 18 months follow-up and signing the consent form.

Exclusion Criteria:

* Patients do not agree the CAD-CAM technique for denture manufacturing.
* Patients refusing participation in the study and signing consent form.
* Patients not willing removable dental restorations.
* Patients not willing to participate at 18 months follow-up evaluation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fully edentulous patients: maxillary, mandible or both dental arches.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of changes in Oral Health Impact Profile for Edentulous Patients (OHIP-EDENT) | up to 18 months
  OHIP-EDENT-RO, validated for Romanian language questionnaire will be administrated at denture insertion and at 6, 12, 18 month follow-up

SECONDARY OUTCOMES:
Evaluation of changes in masticatory performances assessed with Visual Analogue Scale (VAS) | up to 18 months
  At 6, 12 and 18 months clinical follow-up masticatory performance will be evaluated using VAS with units from 0 to 10 where 0 is "totally satisfied" and 10 is "not at all satisfied".
Evaluation of changes in denture retention with VAS | up to 18 months
  At 6, 12 and 18 months denture retention will be evaluated using VAS with units from 0 to 10 where 0 is "strong retention" ("totally satisfied") and 10 is "poor retention"("not at all satisfied").
Evaluation of denture changes in aesthetic aspect with VAS | up to 18 months
  At 6, 12 and 18 months denture aesthetic will be evaluated using VAS with units from 0 to 10 where 0 is "totally satisfied" and 10 is "not at all satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Eftimie Totu, Prof., Study Director — UNIV. POLITEHNICA OF BUCHAREST
Locations (1):
- "Carol Davila"University of Medicine and Pharmacy, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Y, Wen C, Hodgson P, Li Y. Biocompatibility of TiO2 nanotubes with different topographies. J Biomed Mater Res A. 2014 Mar;102(3):743-51. doi: 10.1002/jbm.a.34738. Epub 2013 Jun 1. PMID 23554372
- [Background] Mallineni SK, Nuvvula S, Matinlinna JP, Yiu CK, King NM. Biocompatibility of various dental materials in contemporary dentistry: a narrative insight. J Investig Clin Dent. 2013 Feb;4(1):9-19. doi: 10.1111/j.2041-1626.2012.00140.x. Epub 2012 Dec 17. PMID 23255468
- [Background] Kummer KM, Taylor EN, Durmas NG, Tarquinio KM, Ercan B, Webster TJ. Effects of different sterilization techniques and varying anodized TiO(2) nanotube dimensions on bacteria growth. J Biomed Mater Res B Appl Biomater. 2013 Jul;101(5):677-88. doi: 10.1002/jbm.b.32870. Epub 2013 Jan 29. PMID 23359494
- [Background] Kane RJ, Yue W, Mason JJ, Roeder RK. Improved fatigue life of acrylic bone cements reinforced with zirconia fibers. J Mech Behav Biomed Mater. 2010 Oct;3(7):504-11. doi: 10.1016/j.jmbbm.2010.05.007. Epub 2010 Jun 8. PMID 20696415
- [Background] Gautam R, Singh RD, Sharma VP, Siddhartha R, Chand P, Kumar R. Biocompatibility of polymethylmethacrylate resins used in dentistry. J Biomed Mater Res B Appl Biomater. 2012 Jul;100(5):1444-50. doi: 10.1002/jbm.b.32673. Epub 2012 Mar 27. PMID 22454327
- [Background] Tsuji M, Ueda T, Sawaki K, Kawaguchi M, Sakurai K. Biocompatibility of a titanium dioxide-coating method for denture base acrylic resin. Gerodontology. 2016 Dec;33(4):539-544. doi: 10.1111/ger.12204. Epub 2015 Jul 30. PMID 26223290
- [Result] Totu EE, Nechifor AC, Nechifor G, Aboul-Enein HY, Cristache CM. Poly(methyl methacrylate) with TiO2 nanoparticles inclusion for stereolitographic complete denture manufacturing - the fututre in dental care for elderly edentulous patients? J Dent. 2017 Apr;59:68-77. doi: 10.1016/j.jdent.2017.02.012. Epub 2017 Feb 20. PMID 28223199
- See also: Link to the PRIDENTPRO project. — http://pridentpro.ro/